CLINICAL TRIAL: NCT00006429
Title: Locomotor Therapy Trial for Spinal Cord Injury
Brief Title: Treadmill Training for Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: NICHD-0103; U01HD037439 (NIH)
Record Dates: First submitted 2000-11-01; First posted 2000-11-02 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2011-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Body Weight Supported Ambulation Training; Treadmill Training; Physical therapy; Gait; Assisted Ambulation
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Procedure: body weight-supported treadmill training

SUMMARY:
This is a trial to test whether treadmill training can be used to improve the "walking" of patients with partial spinal cord injury. While on the treadmill, patients will be partially supported through the use of a specially designed harness attached to an overhead lift (also called Body Weight Supported Treadmill Training, BWSTT). Patients who enroll in this study will be randomly assigned to either the experimental group, which receives 12 weeks of this specialized treadmill training with regular physical therapy, or to the control group, which receives 12 weeks regular physical therapy. The ability of the patients to "walk" will be measured before and after treatment as well as 6 and 12 months later, using standard tests that examine mobility independence and speed of ambulation. The trial takes place across five sites in the US and Canada. Patients eligible for this trial will have had a traumatic spinal cord injury within 8 weeks of trial entry.

DETAILED DESCRIPTION:
This is a 5-site randomized clinical trial of a task-oriented locomotor intervention for acute spinal cord injury (SCI). The intervention, body weight-supported treadmill training (BWSTT), partially supports the weight of the patient via an overhead lift attached to a harness. Therapists train the patient to walk on a treadmill by correcting gait deviations and manipulating sensory input that enhance control of the stance and swing phases of walking at increasingly higher speeds and less weight support. 100 patients with incomplete SCI (from below C4 to T10/11) and 100 patients with lesions at T12 to L3 will be randomly assigned to 12 weeks of conventional therapy programs for mobility versus the same intensity and duration of a combination of conventional therapy plus BWSTT. The primary outcome measures are the level of independence for ambulation and the maximal speed for walking 50 feet. Patients will be tested by masked examiners before and after the 12 weeks of therapy, and 6 and 12 months after entry into the study.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury (within 56 days)
* Incomplete lesion: - ASIA C or D, from below C4 to L3 - ASIA B at or below C7
* Unable to ambulate over ground without at least moderate assistance (FIM locomotor 3 or less)
* Able to offer at least 3/5 strength in elbow extensors
* No clinically-significant cognitive impairment

Exclusion Criteria:

* Symptomatic fall in blood pressure greater than 30 mm Hg when upright
* Halo or other cervical brace or TLSO (unless primary surgeon agrees)
* Contraindication to weight bearing on lower extremities
* Pressure sore with any skin breakdown below level of the SCI
* Any debilitating disease prior to the acute SCI that would cause exercise intolerance
* Premorbid, ongoing major depression or psychosis
* Required use of anti-spasticity medication
* Subject unlikely to complete intervention or return for follow-up

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1999-03; Primary Completion 2004-02 (Actual); Study Completion 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H. Dobkin, MD, Principal Investigator — University of California at Los Angeles (UCLA)
Locations (7):
- United States (5):
  - Rancho Los Amigos Medical Center, Downey, California
  - Shepherd Center, Atlanta, Georgia
  - Ohio State University, Columbus, Ohio
  - Six Franklin Plaza, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- Canada (2):
  - University of Ottawa, Ottawa, Ontario
  - McGill University, Montreal, Quebec

REFERENCES:
- [Background] Dobkin, B. "Recovery of Locomotor Control". The Neurologist 1996:239-249.
- [Background] Dobkin, B. "An Overview of Treadmill Locomotor Training with Patrial Body Weight Support: A Neurologically Sound Approach Whose Time Has Come for Randomized Clinical Trials," Neurorehabilitation and Neuronal Repair, 1999 13(3):157-165.
- [Background] Dobkin BH, Apple D, Barbeau H, Basso M, Behrman A, Deforge D, Ditunno J, Dudley G, Elashoff R, Fugate L, Harkema S, Saulino M, Scott M. Methods for a randomized trial of weight-supported treadmill training versus conventional training for walking during inpatient rehabilitation after incomplete traumatic spinal cord injury. Neurorehabil Neural Repair. 2003 Sep;17(3):153-67. doi: 10.1177/0888439003255508. PMID 14503436